CLINICAL TRIAL: NCT07273955
Title: Alcohol Use Disorder Before and After Bariatric Surgery and the Impact of Considering This Surgery During Addiction Follow-up
Acronym: DAACBC
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9372
Record Dates: First submitted 2025-03-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Use Disorder
Keywords: Alcohol Use Disorder; Bariatric Surgery; Alcohol Addiction
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A significant number of patients treated for alcohol use disorder have undergone bariatric surgery.

Bariatric surgery is a treatment for patients suffering from morbid or severe obesity with comorbidities that can be improved by surgery. It is performed by a multidisciplinary team, in collaboration with the treating physician. It is a comprehensive approach, part of a personalized patient plan, and is governed by regulations defined by the HAS (French National Authority for Health). Pre- and post-surgery follow-up are defined within these regulations.

Several studies have been conducted on alcohol use disorder after bariatric surgery, attempting to understand and clarify the mechanisms involved. Alcohol use disorder and bariatric surgery share and are associated with psychiatric disorders.

Therefore, the investigators wish to explore, through the medical records of patients receiving addiction treatment for alcohol use disorder, the consideration of their surgery in their follow-up. This exploration will subsequently allow for improved care for these patients, if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Adult (≥18 years old)
* Female or male
* Having undergone bariatric surgery
* History of eating disorders before or after bariatric surgery
* History of AUD before or after bariatric surgery
* Other substance use disorder
* Addiction follow-up at the CSAPA of the HUS or Saverne hospitals for an alcohol use disorder during the period from January 1, 2003 to March 31, 2024
* Subject not objecting, after being informed, to the reuse of their data for the purposes of this research

Exclusion Criteria:

* Patient who has expressed opposition to participating in the study.
* Absence of alcohol use disorder. - No bariatric surgery.
* Patient under legal protection, guardianship, or curatorship.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult (≥18 years old) having undergone bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2025-12-12 (Estimated); Study Completion 2025-12-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients suffering from eating disorders and alcohol use before and after bariatric surgery, over the period from January 1, 2003 to March 31, 2024. | Up to 1 year after bariatric surgery

CONTACTS AND LOCATIONS:
Locations (1):
- (Centre de Soins, d'accompagnement et de prévention en Addictologie - CHU de Strasbourg - France, Strasbourg, France